CLINICAL TRIAL: NCT06416332
Title: Development and Implementation of a Tele -Rehabilitation System for Patients With Knee Osteoarthritis (Aged 40-70 Years, Kellgren Grade 1-3 and Lawrence )
Brief Title: Development and Testing of a Tele-rehabilitation System for Adult Patients With Knee Osteoarthritis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of West Attica (Other)
Responsible Party: Principal Investigator, Theodora Plavoukou, PT,MSc,PhD(can)Physiotherapy Department of the University West Attica, University of West Attica
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 61123-27/06/2023
Record Dates: First submitted 2024-05-07; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Knee Osteoarthritis; Knee Osteoarthritis (OA); Telerehabilitation
Keywords: Exercise; knee osteoarthitis; tele-rehabilitation; physical therapy
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
  This a randomized controlled trial with first primary end point at 8 weeks and second primary end point at 3 months. Participants will be allocated randomly into one of two intervention groups. Group1 (Telerehabilitation) Group 2 (in person)
Who Masked: Investigator, Outcomes Assessor
Masking Description: The Investigator and outcomes assessor are blinded to patient allocation and data code.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- in face to face live group (Experimental): In the live therapeutic exercise group (group A) the program and its progression will be determined and performed for life according to the patient's progress, with a frequency of sessions twice a week, a session duration of 45 minutes, following the recommended dosage of exercise according to with the clinical instructions, while the total duration of the intervention will be eight weeks.
  Interventions: Other: group A: in face to face live therapeutic exercise
- telerehabilitation program group (Experimental): In the telerehabilitation program group (group B), the therapeutic exercise program will follow the same structure, with differences in the explanation of the exercises, their presentation, as well as the monitoring and information of the participants, as they will be done through a telerehabilitation platform and a special software data processing. The intervention time remains the same, with the physiotherapist in these 45 minutes of the session evaluating the data on the patient's progress by receiving the information through the software, and informing the patient of any changes in the progression of the exercise program. The remaining parameters of the intervention also remain the same, as in face to face live exercise.
  Interventions: Other: group B: telerehabilitation program

INTERVENTIONS:
Other: group A: in face to face live therapeutic exercise — In group A: in face to face live therapeutic exercise the program and its progressivity will be determined and performed for life according to the progress of the patient, with a frequency of sessions twice a week, session duration 45 minutes, following the recommended dosage of exercise according to clinical guidelines, while the total duration of the intervention will be eight weeks. You will be instructed to perform the program at home, 3 times a week. The standardized exercise program to be followed by this group will include :
  1. Exercises to strengthen the hip and knee muscles through isometric contractions and resistance exercises using elastic bands.
  2. Balance and neuromuscular coordination exercises.
  Arms: in face to face live group
Other: group B: telerehabilitation program — In group B: telerehabilitation program, the therapeutic exercise program will follow the same structure, which was mentioned above. The differentiation in the intervention of this group will be that the explanation of the exercises, their presentation, monitoring and information of the participants will be done through the telerehabilitation platform and special data processing software. The intervention time remains the same, with the physical therapist during these 45 minutes of the session , to evaluate the data on the patients progress by receiving the information through the software and to inform the patient of any changes in the progressivity of the exercise program. The other parameters of the intervention remain the same, as in person exercise.
  Arms: telerehabilitation program group

SUMMARY:
DEVELOPMENT AND TESTING OF A TELEREHABILITION SYSTEM FOR PATIENTS WITH OSTEOARTHRITIS OF THE. KNEE (AGES 40-70 YEARS, GRADE 1-3, ACCORDING TO KELLGREN AND LAWRENCE) This study aims to develop and compare two methods of implementing a therapeutic exercise program for knee osteoarthritis: face-to-face sessions versus a telerehabilitation program. The telerehabilitation system will allow remote delivery of exercises with real-time monitoring and feedback. Measurement tools will assess various dimensions of knee osteoarthritis, ensuring comprehensive evaluation. Two experimental groups will receive either face-to-face or telerehabilitation sessions twice a week for eight weeks. Both groups will follow structured exercise programs, with the telerehabilitation group receiving remote instructions and feedback. Measurements will be taken before and after the intervention period, as well as at a three-month follow-up. Expected results include confirming and potentially enhancing findings regarding the effectiveness of remote rehabilitation for knee osteoarthritis. The study anticipates that telerehabilitation intervention could be equally or more effective than face-to-face intervention, ultimately providing a personalized, self-managed solution for managing chronic conditions like knee osteoarthritis.

DETAILED DESCRIPTION:
The purpose of this study is to develop, investigate and compare the effectiveness of a new system of remote therapeutic exercise, using technological equipment, in relation to face to face therapeutic exercise, which is proposed by international guidelines, in patients with osteoarthritis of the knee. More specifically, the magnitude of the improvement of motor, kinematic and psychocognitive parameters, physical condition, functionality, quality of life and symptoms of the disease will be examined, using these two methods. It is fully understood and constitutes one of the objectives of this study , that the volume of this information should be transmitted to the patient and the physical therapist in the most understandable and simplified way possible. Finally, the effectiveness of the interventions will also be evaluated in relation to the ease of use and execution of the therapeutic exercise plan, as well as the degree of compliance of the patients with each intervention method.

The aim of the present study is the development of an innovative telerehabilitation system and the comparison of two different methods of implementation of a therapeutic exercise program for knee osteoarthritis, and in particular a face to face live program and a remote application program. In order to implement remote intervention, a rehabilitation system for patients with knee osteoarthritis will be created, where therapeutic exercise will be provided through special software and technological equipment and the patients progress will be monitored remotely or in real time, whenever this is deemed necessary. . In this way, it is expected to create a remote but immediate rehabilitation environment, with easy access, which will provide flexibility, short response time and economy during its application by the patient.

This study is a multicenter, single-blind, randomized, controlled prospective study with two parallel axes will be designed. The sample will come from the places where the study will be carried out and which are legal physical therapy laboratories.The participants of this study will be volunteers a considedered a sample of men and women, aged 40-70 years with radiographically and orthopedically diagnosed knee osteoarthritis, Kellgren grade 1-3 and Lawrence classification system of osteoarthritis.

The Sample size was determined by the G- power test analysis based on the primary outcome measures selected and the effect size size which is reported in similar studies. According to a meta-analysis, the effect size for pain measures ( whether the measurements were made using questionnaires or algometers ) was equal to SMD =0.66, in all the measurement tools used . Finally, in a research, in which the isokinetic dynamometer was used as a measuring tool, the effect size for the strength of the subjects quadriceps muscle was equal to SMD =0.42. Thus, taking into account all the above and setting the level of statistical significance at α=0.05 and the power of the study at 80%, through the G- power analysis test the sample size was determined at 34 participants. Assuming a potential loss to follow-up of 20% of participants, the minimum sample size was calculated at 42 patients.

The randomization process will be performed by an independent researcher. The allocation of participants will be done randomly through the use of the random.org program. Sealed envelopes will be given to participants prior to their allocation to research groups and each envelope will indicate the group to which each participant is allocated, as randomly assigned by the computer program.

The study will have two experimental groups , group A : face to face therapeutic exercise and group B: telerehabilitation program.

In group A: for face to face live therapeutic exercise the program and its progressivity will be determined and performed face to face according to the progress of the patient, with a frequency of sessions twice a week, session duration 45 minutes, following the recommended dosage of exercise according to clinical guidelines, while the total duration of the intervention will be eight weeks. You will be instructed to perform the program at home, 3 times a week. The standardized exercise program to be followed by this group will include :

1. Exercises to strengthen the hip and knee muscles through isometric contractions and resistance exercises using elastic bands.
2. Balance and neuromuscular coordination exercises. This standardized program will be structured following international guidelines and the gradual difficulty of the exercises will be confirmed through electromyographic activity of the respective muscle groups, following a pilot study, the results of which will be the mechanism for confirming the progression of the difficulty of each exercise, so that the patient can either proceed according to his progress to the next exercise, or return to a previous exercise if he experiences pain during its execution.

Initially, patients will be informed about the pathogenesis and the proposed, according to the article, management of the disease. Then, there will be a documentation and explanation of the progressive therapeutic exercise program, as suggested by the international literature, while printed material will also be distributed.

In group B: telerehabilitation program, the therapeutic exercise program will follow the same structure, which was mentioned above. The differentiation in the intervention of this group will be that the explanation of the exercises, their presentation, monitoring and information of the participants will be done through the telerehabilitation platform and special data processing software, as shown in diagram 1. The intervention time remains the same, with the physical therapist during these 45 minutes of the session , to evaluate the data on the patients progress by receiving the information through the software and to inform the patient of any changes in the progressivity of the exercise program. The other parameters of the intervention remain the same, as in the face to face live exercise.

All participants will initially complete a questionnaire that will include their history and demographics. They will complete the study questionnaires and submit to the respective tests, the same procedure will be followed after the eight weeks and the end of the respective interventions in both intervention groups and the same procedure will be followed after the three months.

The statistical processing will be done with SPSS (Statistical Package for the Social Science) software for Windows (version 25.0). A statistical analysis will be performed of the differences of each measurement, between the two interventions, as they will be recorded before the start of the intervention, eight weeks and three months later, using the MANOVA and Kruskal - Wallis test (for the non-parametric data). Data normality testing will be performed and the statistical significance level will be set at α = 0.05.

With the completion of this research work, it is expected to confirm and increase the findings of previous studies in the international literature regarding the effect of remote rehabilitation through an innovative telerehabilitation system, for patients suffering from knee osteoarthritis, through a series of assessment tools that do not have so far been described in combination. Evidence is awaited that telerehabilitation intervention will be equally - or even more - effective than in-person intervention. The ultimate and final goal will be to create an optimal, personalized environment for self-management of such a chronic pathological entity as knee osteoarthritis, with the perspective that this intervention will be the optimal solution for managing chronic diseases .

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-70
2. Ability to provide consent and good knowledge of the Greek language
3. Diagnosed, radiographically and by an orthopedic doctor, knee osteoarthritis grade 1-3, according to Kellgren and Lawrence classification system of osteoarthritis
4. Diagnosis of knee osteoarthritis and good general health

Exclusion Criteria:

1. Participation in a systematic exercise program in the previous three months for the same problem
2. Participation in a physical therapy program in the previous three months for the same problem
3. Previous knee surgery within last three years
4. Medical contraindication to exercise
5. Systemic diseases or autoimmune in the acute phase of symptoms
6. Underlying severe neurological disease
7. Cognitive disability → inability to communicate
8. Red Flags (eg fractures (osteoporotic and non-osteoporotic), rapidly unexplained decrease in muscle strength, cardiorespiratory problems, etc.)

   -

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
pain and stiffness of the knee joint | [Time Frame: baseline, 8 weeks (end of treatment), 3 months (follow up)]
  "change" is being assessed for pain and stiffness of the knee joint with The WOMAC tool (Western Ontario and McMasters Universities Osteoarthritis Index), is a widely used measure. The questionnaire consists of 24 sections which are divided into three subscales . A five-point Likert (0-4) isosceles scale is used for calibration . Thus the pain subscale can be scored from 0-20, the stiffness 0-8 and the functionality 0-68. In addition to the Linkert scale, the VAS scale (visual analog scale) can be used. On a straight line of 10 cm, from 0 (no pain) to 10 (worst pain), the patient notes the pain he is experiencing at that moment. The WOMAC questionnaire is reliable and valid, the Greek version has been checked for its validity and reliability in a research.
the muscle performance of the quadriceps muscle | [Time Frame: baseline, 8 weeks (end of treatment), 3 months (follow up)]
  "change" is being assessed for the muscle perfomance done with the help of the surface electromyogram with and the use of an isokinetic dynamometer, which are also considered as the gold standard standard .

SECONDARY OUTCOMES:
functionality | Time Frame: baseline, 8 weeks (end of treatment), 3 months (follow up)]
  "change" is being assessed for functionality with ASES.The Arthritis Self-Efficacy Scale (ASES) was developed to explain changes in the health of arthritis patients following educational interventions. KAA (Arthritis Self-Efficacy Scale - ASES) is the most frequently used and psychometrically tested tool specialized in arthritis. The KAA is a tool for assessing self -efficacy in patients with arthritis . The KAA includes 20 questions that assess three (3) factors: a) Pain self -efficacy - AP (5 questions), b) Functionality self-efficacy - AL (9 questions) and c) Other Symptoms self-efficacy - AAS (6 questions). Question scores range from 1 (not at all sure) to 10 (very sure) on a numerical scale, with continuous vertical lines representing whole numbers. The score of each factor results from the average of its individual questions. The scale should not be scored if more than 25% of the total questions have not been answered. The time to complete the KAA is estimated at 5-10 minutes.
Kinesiophobia | Time Frame: baseline, 8 weeks (end of treatment), 3 months (follow up)
  "change" is being assessed for Kinesiophobia with TSK.The TSK scale is a widely used tool that measures fear of movement or re-injury in various activities. It consists of 17 questions that can take four values from value 1: completely disagree to value 4: completely agree. The total score is calculated after reversing questions 4, 8, 12 and 16. The Greek version of the Tampa scale Scale of Kinesiophobia was measured in Greek and the validity and reliability indices of the Greek version were examined by the study , where they demonstrated a valid and reliable assessment tool whose internal validity (Cronbach's a=0.74) and reliability (ICC=0.78) demonstrate a tool capable of measuring patients' perception of fear of re-injury due to exercise or physical activity.
Balance - Propriety | Time Frame: baseline, 8 weeks (end of treatment), 3 months (follow up)]
  "change" is being assessed for Balance - Propriety is Time Up and Go Test .Time up and Go test: introduced in 1991 by Podsiadlo and Richarson as a measure of physical performance. Requires minimal equipment. The patient is asked to get up from a chair 45-50 cm high without sides, come to a standing position, travel as fast as possible a distance of three meters, turn and return to his original position. The total time of the test is related to the patient's level of functional ability.
Anxiety - Depression | Time Frame: baseline, 8 weeks (end of treatment), 3 months (follow up)]
  for Anxiety - Depression is the Hospital Anxiety and Depression Scale (HADs) The Hospital Anxiety and Depression Scale (HADs): The HADs tool is a self-reported and calibrated scale measuring anxiety and depression. This scale consists of 14 questions, with a range of values from 0 to 3, which are divided into two subcategories. One subscale includes seven questions to screen for depression and the other with the same number of questions screens for anxiety disorders. The sum of the representative questions for each disease (0-21) forms an attempt to highlight the severity and quantification of anxiety and depression. The Hospital Anxiety and Depression Scale (HADS) is used to study anxiety and depression in hospital patients . The scale is completed by the examinee himself and consists of a total of 14 questions. Specifically, two factors are studied, anxiety (HADS-Anxiety - HADS-A) and depression (HADS-Depression - HADS-D), with each factor including 7 questions.
Compliance | Time Frame: baseline, 8 weeks (end of treatment), 3 months (follow up)]
  change" is being assessed for Compliance with Diary of continuous recording of exercise time either in physical form or online

CONTACTS AND LOCATIONS:
Overall Officials: Theodora Plavoukou, PhDc, Principal Investigator — uniwa; George Georgoudis, PhD, Study Director — uniwa
Locations (1):
- Physiotherapy Department, University of West Attica, Athens, Agiou Spiridonos 28, 12243 Egaleo,, Greece

IPD SHARING:
Plan to Share IPD: Yes
Yes
  Only upon agreement by the authors that there will be no further changes and/ or analysis, results of the study will be published and shared. No patient data will be shared to be compliant with the latest GDPR code.
Supporting Information: Study Protocol, CSR
Time Frame: 6 months after publication date and only upon agreement by the authors that there will be no further changes and/or analysis may data be shared.
Access Criteria: It is to the authors discretion to share study data to other researchers.

REFERENCES:
- [Background] Skrepnik N, Spitzer A, Altman R, Hoekstra J, Stewart J, Toselli R. Assessing the Impact of a Novel Smartphone Application Compared With Standard Follow-Up on Mobility of Patients With Knee Osteoarthritis Following Treatment With Hylan G-F 20: A Randomized Controlled Trial. JMIR Mhealth Uhealth. 2017 May 9;5(5):e64. doi: 10.2196/mhealth.7179. PMID 28487266
- [Background] Saki, F., Bakhtiari Khou, S. and Ramezan, F. (2020). The Role of Digital Technologies as an Alternative for Face-to-Face Knee Rehabilitation: A Systematic Review. Physical Treatments: Specific Physical Therapy Journal, 10(4), pp.185-194
- [Background] Naeemabadi, Mr., Fazlali, H., Najafi, S., Dinesen, B. and Hansen, J. (2020). Telerehabilitation for Patients With Knee Osteoarthritis: A Focused Review of Technologies and Teleservices. JMIR Biomedical Engineering, 5(1), p.e16991.
- [Background] Mecklenburg G, Smittenaar P, Erhart-Hledik JC, Perez DA, Hunter S. Effects of a 12-Week Digital Care Program for Chronic Knee Pain on Pain, Mobility, and Surgery Risk: Randomized Controlled Trial. J Med Internet Res. 2018 Apr 25;20(4):e156. doi: 10.2196/jmir.9667. PMID 29695370
- [Background] Kolasinski SL, Neogi T, Hochberg MC, Oatis C, Guyatt G, Block J, Callahan L, Copenhaver C, Dodge C, Felson D, Gellar K, Harvey WF, Hawker G, Herzig E, Kwoh CK, Nelson AE, Samuels J, Scanzello C, White D, Wise B, Altman RD, DiRenzo D, Fontanarosa J, Giradi G, Ishimori M, Misra D, Shah AA, Shmagel AK, Thoma LM, Turgunbaev M, Turner AS, Reston J. 2019 American College of Rheumatology/Arthritis Foundation Guideline for the Management of Osteoarthritis of the Hand, Hip, and Knee. Arthritis Rheumatol. 2020 Feb;72(2):220-233. doi: 10.1002/art.41142. Epub 2020 Jan 6. PMID 31908163
- [Background] Johnson AJ, Palit S, Terry EL, Thompson OJ, Powell-Roach K, Dyal BW, Ansell M, Booker SQ. Managing osteoarthritis pain with smart technology: a narrative review. Rheumatol Adv Pract. 2021 Mar 16;5(1):rkab021. doi: 10.1093/rap/rkab021. eCollection 2021. PMID 33928214
- [Background] Byra J, Czernicki K. The Effectiveness of Virtual Reality Rehabilitation in Patients with Knee and Hip Osteoarthritis. J Clin Med. 2020 Aug 14;9(8):2639. doi: 10.3390/jcm9082639. PMID 32823832
- [Background] Bennell K, Nelligan RK, Schwartz S, Kasza J, Kimp A, Crofts SJ, Hinman RS. Behavior Change Text Messages for Home Exercise Adherence in Knee Osteoarthritis: Randomized Trial. J Med Internet Res. 2020 Sep 28;22(9):e21749. doi: 10.2196/21749. PMID 32985994
- [Background] Allen KD, Arbeeva L, Callahan LF, Golightly YM, Goode AP, Heiderscheit BC, Huffman KM, Severson HH, Schwartz TA. Physical therapy vs internet-based exercise training for patients with knee osteoarthritis: results of a randomized controlled trial. Osteoarthritis Cartilage. 2018 Mar;26(3):383-396. doi: 10.1016/j.joca.2017.12.008. Epub 2018 Jan 5. PMID 29307722
- [Derived] Plavoukou T, Kasnesis P, Contiero Syropoulou A, Papagiannis G, Stasinopoulos D, Georgoudis G. A Sensor-Augmented Telerehabilitation System for Knee Osteoarthritis: A Randomized Controlled Trial of Neuromuscular, Functional, and Psychosocial Outcomes. Sensors (Basel). 2025 Nov 21;25(23):7113. doi: 10.3390/s25237113. PMID 41374487